CLINICAL TRIAL: NCT05964868
Title: The Efficacy of Liposomal Bupivacaine in the Management of Post-operative Pain Following Septorhinoplasty: a Single-blinded, Prospective Clinical Trial
Brief Title: Efficacy of Liposomal Bupivacaine Post Septorhinoplasty
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Jessyka Lighthall (Other)
Responsible Party: Sponsor-Investigator, Jessyka Lighthall, Chief, Division of Facial Plastic & Reconstructive Surgery, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00020710
Record Dates: First submitted 2023-07-06; First posted 2023-07-28 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Rhinoplasty; Pain Management
Keywords: Narcotics; opioid; septorhinoplasty; pain
MeSH Terms: conditions — Agnosia; Pain | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled, single-blinded study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient, surgeons, and research team will be blinded to the group that the subject was randomized to. The pharmacy will prepare equivalent drugs for each study group to visually appear similar so that blinding can be maintained. In the event if the patient experiences a concerning or an adverse reaction, the patient, the surgeons and the research team will be immediately unblinded from the study. If unblinding is required, the pharmacy will be notified and then will provide, from the randomization list, information as to which study group the patient was assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Liposomal Bupivacaine (Experimental): This group will receive a one time 5 mL injection of liposomal bupivacaine post-operatively at the surgical site.
  Interventions: Drug: Liposomal Bupivacaine
- Bupivacaine with epinephrine (Active Comparator): This group will receive a one-time 5 mL injection of 0.25% bupivacaine with 1:200,000 epinephrine post-operatively at the surgical site.
  Interventions: Drug: 0.25% bupivacaine with 1:200,000 epinephrine
- Saline solution (Placebo Comparator): This group will receive a one-time 5 mL injection of saline post-operatively at the surgical site.
  Interventions: Other: Placebo - Saline solution

INTERVENTIONS:
Drug: Liposomal Bupivacaine — Patients will receive post-operative liposomal bupivacaine (EXPAREL®) at the surgical site at the completion of their septorhinoplasty.
  Arms: Liposomal Bupivacaine
Drug: 0.25% bupivacaine with 1:200,000 epinephrine — Non-liposomal encapsulated bupivacaine at the surgical site at the completion of septorhinoplasty.
  Arms: Bupivacaine with epinephrine
Other: Placebo - Saline solution — This group will receive a one-time 5 mL injection of saline post-operatively at the surgical site.
  Arms: Saline solution

SUMMARY:
The objective of this study is to determine if there is a difference in post-operative pain after septorhinoplasty when long-acting liposomal bupivacaine is used for local anesthesia compared to other standard local anesthetic regimens.

DETAILED DESCRIPTION:
Hypothesis: Patients receiving postoperative liposomal bupivacaine (EXPAREL®) at the surgical site after their septorhinoplasty will have better postoperative pain control and require fewer narcotics by means of a lower MME compared to the placebo group and the group that receives postoperative 0.25% bupivacaine with 1:200,000 epinephrine.

This a prospective randomized controlled, single-blind study evaluating the efficacy of EXPAREL® versus plain bupivacaine HCl and placebo after perinasal injections during septorhinoplasty procedures. Seventy-two total patients undergoing septorhinoplasty will be randomly distributed into three groups (20 patients per group) with various postoperative local anesthesia regimens. All groups will be given standard oral postoperative pain regimens as prescribed by the primary surgeon, typically consisting of alternating doses of 1000 mg acetaminophen and 800 mg ibuprofen with oxycodone 5 mg every 6 hours as needed for breakthrough pain. All three groups will receive the same treatment at the beginning of surgery with pre-incisional local surgical site injections with perinasal blocks of 1% lidocaine with 1:100,000 epinephrine. Group one (study group) will receive a five mL injection of EXPAREL® postoperatively, group two will receive a five mL injection of 0.25% bupivacaine with 1:200,000 epinephrine postoperatively, and group three will receive a five mL injection of saline along the surgical site, all in a ring block fashion (see illustration). This ring block involves nerve blocks to nasal branches of the supratrochlear, infraorbital, and infratrochlear nerves. This will also be injected into the floor of the nasal cavity to block branches of the nasopalatine nerve. The remainder of the ring block targets local infiltration surrounding the nose and injections are over bone. Although there is a potential risk of diffusion to adjacent cartilage, this risk is predicted to be low. Their use of postoperative pain medications will then be documented in the immediate postoperative period in the post-anesthesia care unit (PACU) as well as the following week postoperatively, every day, for three times a day. All groups will be required to fill electronic pain journals through RedCap (a HIPPA compliant server) to record consumption of pain medications and pain levels as reported by visual analog pain scales, the Wong-Baker FACES pain rating scale, and modified McGill pain questionnaire, all of which are validated tools for pain assessment. Patients will be subsequently followed over the course of six months postoperatively with these validated measures, use of pain medication, and by clinical exam of the nose/injection site including both external and internal nasal exam, palpation of the nose and cartilage grafts, evaluation static and dynamic function of the nose, and the presence of any adverse outcomes including but not limited to cartilage graft loss, septal perforation, synechiae formation, infection, and persistent or worsening nasal obstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be undergoing rhinoplasty or septorhinoplasty surgery
2. Male or female subjects greater than or equal to 18 years of age
3. Written informed consent must be obtained

Exclusion Criteria:

2. The subject is a pregnant or lactating 3. Patients have a cognitive impairment 4. Patient is a prisoner 5. Patients with hypersensitivity to local anesthetics and pain medications used in the study 6. Patients weighing less than 48 kg 7. Patients preoperatively taking narcotics for chronic pain 8. Patients with pre-existing painful conditions (complex regional pain syndrome, fibromyalgia, neuropathy) 9. Patients with liver dysfunction 10. Patients with increased creatinine (over 1.5 mg/dl) 11. Patients who have undergone autologous costal cartilage grafting with their rhinoplasty 12. Morbid obesity (BMI >40)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Differences in postoperative milligram morphine equivalents (MME) used between placebo and liposomal bupivacaine | 6 months
  Convert amount of opioid ingested to MMEs as an objective measure of post-operative narcotic use

SECONDARY OUTCOMES:
Different in patient reported outcome measure of subjective pain scores based on a validated visual analog pain scale (subjective measure) between placebo and test drug | 6 months
  Validated universal pain assessment tool: Wong-Baker pain scale pain questionnaire. Min 0 = no pain to 10 = maximum pain
Difference in time to first dose of opioid rescue after surgery between placebo and test drug | 6 months
  measure the time from leaving surgery to when the first dose of opioid is taken
Difference in breathing outcomes between placebo and test drug | 6 months
  NOSE questionnaire minimum 0 no obstruction to 100 complete obstruction
Difference in adverse events/complications between placebo and test drug | 6 months
  Assess for general adverse events and post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Jessyka Lighthall, MD, Principal Investigator — Penn State Health
Locations (1):
- Jessyka Lighthall, Hershey, Pennsylvania, United States